CLINICAL TRIAL: NCT06948695
Title: Evaluation of the Biomechanics of Crowding and the Energetic Cost of Endurance Runners Unilateral Transtibial Amputees According to the Stiffness of the Race-specific Prothesis.
Brief Title: Evaluation of the Biomechanics of Crowding and the Energetic Cost of Endurance Runners Unilateral Transtibial Amputees.
Acronym: BLADENDURUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24CH148; 2024-A01795-42 (Other: ID RCB)
Record Dates: First submitted 2025-02-07; First posted 2025-04-29 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Amputee; Prostheses; Healthy Volunteers
Keywords: Unilateral transtibial amputees; Endurance runners
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: prospective randomized cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual blade stiffness (Active Comparator): Data collection on a blade with usual stiffness during a run at comfort speed according to slope (flat, uphill +10% and downhill -10% on treadmill) and type of terrain (road, path).
  Interventions: Other: Warm-up; Other: Random blade test; Other: Comfort speed test; Other: Outdoor random blade test
- Less stiff blade (Active Comparator): Data collection on a less stiff blade during a run at comfort speed according to slope (flat, uphill +10% and downhill -10% on treadmill) and type of terrain (road, path).
  Interventions: Other: Warm-up; Other: Random blade test; Other: Comfort speed test; Other: Outdoor random blade test
- Stiffer blade (Active Comparator): Data collection on a stiffer blade during a run at comfort speed according to slope (flat, uphill +10% and downhill -10% on treadmill) and type of terrain (road, path).
  Interventions: Other: Warm-up; Other: Random blade test; Other: Comfort speed test; Other: Outdoor random blade test

INTERVENTIONS:
Other: Warm-up — 5-minute warm-up run on treadmill at a freely chosen speed
Other: Random blade test — 4-minute run on a treadmill with a flat incline.
Other: Random blade test — 4-minute run on treadmill with a 10% gradient
Other: Comfort speed test — 1 min running test on an instrumented treadmill (Gaitway, H/P/Cosmos, Nußdorf, Germany) at comfort speed.
Other: Outdoor random blade test — 100-metre outdoor run at a comfort speed

SUMMARY:
Transtibial amputation accounts for 3,700 cases per year in France. Athletes can use sport blades made of carbon plate for improved energy restitution.

Sports blades are adjusted according to the manufacturer's recommendations and the subjective experience of the ortho-prosthetist and patient. These adjustments are designed to optimize performance and comfort while reducing the risk of injury. This risk is all the greater when asymmetries between the healthy and affected limbs are large, exposing the healthy limb to large and repeated reaction forces.

DETAILED DESCRIPTION:
Furthermore, one of the performance criteria for long-distance running is energy cost. While a reduction in this parameter has been observed in bilateral amputees, heterogeneous data are reported in unilateral amputees, depending on the level of expertise and sports blade settings.

While studies have investigated the effects of running with a prosthesis under conditions representative of track running, few data are available on sports blades designed for long-distance running.

It therefore seems important to be able to objectively assess the effects of a change in the stiffness of the sports blade on the energetics and biomechanics of running, in order to optimize practice and prevent associated traumas.

Secondly, investigators believe it is important to verify that the biomechanical results obtained in the laboratory are applicable in the field, both on the road and on the unstable terrain encountered by trail runners.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Weighing less than 110 kg, in accordance with C-blade recommendations,
* Subjects who have undergone a unilateral transtibial amputation,
* Have been running with a sports blade for at least 3 months, over several sessions of at least 3 kilometers.
* Subjects who have signed a written consent form,
* Subjects affiliated or entitled to a social security scheme.

Exclusion Criteria:

* Subjects whose amputation is due to complications related to diabetes or atherosclerosis.
* Subjects with chronic or central neurological pathologies
* Subjects with cardiovascular disorders
* Subjects with alcohol or drug dependency.
* Pregnant or breast-feeding women
* Subjects under court protection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption measurement | Day 1
  4-minute flat run on a treadmill at comfort speed

SECONDARY OUTCOMES:
Oxygen consumption measurement | Day 1
  4-minute up hill run (+10%), on a treadmill at comfort speed
Kinematic analysis | Day 1
  Slope-dependent kinematic analysis by measuring joint angles (in degrees), moments (Nm) and net joint forces at ankle, knee and hip (in Nm/Kg), ground reaction forces (in N/Kg) during a 1-minute run on different slopes (downhill -10%, flat, uphill +10%).
Cadence of running (in steps per minutes) | Day 1
  Cadence of running according to slope (downhill -10%, flat, uphill +10%) and terrain, measured during a 1-minute run on a carpet
Stride length (in meters) of running | Day 1
  Stride length of running according to slope (downhill -10%, flat, uphill +10%) and terrain, measured during a 1-minute run on a carpet
Cadence (in steps per minute) of running | Day 2
  Cadence of running according to gradient (downhill -10%, flat, uphill +10%) and type of terrain, measured during a 100-metre run on roads and paths.
Stride length (in metres) of running | Day 2
  Stride length (in metres)of running according to gradient (downhill -10%, flat, uphill +10%) and type of terrain, measured during a 100-metre run on roads and paths.
Leg muscle activity (mV) | Day 1, 2
  Recording of leg muscle activity under all conditions using surface electromyographic recordings (Trigno wireless electromyogram (EMG) electrodes (Delsys, Natick, USA) made on the vastus lateralis, rectus femoris and gluteus medius muscles (Root Mean Square (RMS).
Subjective sensation recording | Day 1, 2
  Recording of the subjective sensation of perceived exertion at the end of each condition using a Borg scale ranging from 0 to 10.
  0 = It is very very easy 10= so hard that I have to stop

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD-PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: Undecided